CLINICAL TRIAL: NCT06530615
Title: Investigation of Microplastic Pollution in the Human Respiratory System and Its Relationship to Lung Cancer
Brief Title: Investigation of MP Pollution in the Human Respiratory System and Its Relationship to Lung Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: MCC-22605
Record Dates: First submitted 2024-07-26; First posted 2024-07-31 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Lung Cancer
Keywords: Microplastic Pollution; Human Respiratory System
MeSH Terms: conditions — Lung Neoplasms | interventions — Bronchoalveolar Lavage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lung Neoplasm: Lung Cancer cases will be comprised of patients that are confirmed to have lung cancer based on bronchoscopy/ Bronchoalveolar Lavage (BAL) and other clinical testing.
  Interventions: Procedure: Bronchoalveolar Lavage (BAL) during Bronchoscopy
- Lung Neoplasm Excluded: Lung Cancer excluded cases will be comprised of the remaining patients in whom lung cancer is excluded as a diagnosis based on bronchoscopy/ Bronchoalveolar Lavage (BAL) and other clinical testing.
  Interventions: Procedure: Bronchoalveolar Lavage (BAL) during Bronchoscopy

INTERVENTIONS:
Procedure: Bronchoalveolar Lavage (BAL) during Bronchoscopy — Bronchoalveolar Lavage (BAL) is a standard diagnostic tool for the evaluation of lower respiratory tract pathology including respiratory infections and unexplained radiographic pulmonary lesions including lung neoplasia. It is a minimally invasive procedure that involves introduction of the bronchoscope, installation of sterile normal saline into a subsegment of the lung, and suction and collection of the recovered saline for diagnostic evaluation.

SUMMARY:
This project will study and characterize Microplastic (MP) burden in the lungs of patients undergoing Bronchoalveolar Levage (BAL) in thoracic clinics at Moffitt.

ELIGIBILITY:
Inclusion Criteria:

* English or Spanish-speaking patients scheduled for bronchoscopy/bronchoalveolar lavage (BAL) in thoracic clinics at Moffitt.

Exclusion Criteria:

* Patients with a known prior history of lung cancer or that have undergone a Bronchoalveolar Lavage (BAL) procedure at any time in the past in the involved lung targeted for BAL.
* Patients that have had any prior lung or thoracic or surgeries or procedures (examples: removal of lung or portions of the involved lung (lobectomy, pneumonectomy, wedge resection/segmentectomy).
* Patients with specimens that are considered to be non-adequate as true Bronchoalveolar Lavage Fluid (BALF) (i.e., absence of alveolar macrophages) after pathologist's evaluation will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any Moffitt patient undergoing bronchoscopy/bronchoalveolar lavage (BAL) either English or Spanish speaking.
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2024-02-05 (Actual); Primary Completion 2026-09-18 (Estimated); Study Completion 2026-09-18 (Estimated)

PRIMARY OUTCOMES:
Characterization of Microplastic (MP) Burden in the Lungs | Up to 24 Months
  Microplastic (MP) Burden in the Lungs will be determined by the results of the Bronchoscopy/Bronchoalveolar Lavage (BAL).
  MPs isolated from Bronchoalveolar Fluid (BALF) will be characterized using Raman spectroscopy (RS). RS is a vibrational spectroscopy technique based on the inelastic scattering of light that provides information on the molecular vibrations of a system in the form of a vibrational spectrum. The Raman spectrum is akin to a fingerprint of chemical structure allowing identification of the components present in the sample.
  For each sample, data will be generated on the presence or absence of MPs, total number of MPs, and polymer subtype distribution of MPs identified in the samples.

SECONDARY OUTCOMES:
Concentration of Microplastics (MPs) in Lung Cancer Patients | Up to 24 Months
  Concentration of Microplastics (MPs) will be determined by the number of MPs identified in 10-mLs of Bronchoalveolar Fluid (BALF).
Concentration of Microplastics (MPs) in Non-Lung Cancer Patients | Up to 24 Months
  Concentration of Microplastics (MPs) will be determined by the number of MPs identified in 10-mLs of Bronchoalveolar Fluid (BALF).

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen M Egan, ScD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trials Website — http://www.moffitt.org/clinical-trials-research/clinical-trials/